CLINICAL TRIAL: NCT02648386
Title: Bone Marrow Mononuclear Cells or Human Umbilical Cord-derived Mesenchymal Stem Cells Combined With NeuroRegen Scaffold™ Transplantation for the Improvement of Erectile Function in Men After Rectal Cancer Surgery
Brief Title: Stem Cell Therapy Combined With NeuroRegen Scaffold™ in Patients With Erectile Dysfunction After Rectal Cancer Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CAS-XDA-ED-IGDB
Record Dates: First submitted 2016-01-05; First posted 2016-01-07 (Estimated); Last update posted 2019-01-25 (Actual); Status verified 2015-12

CONDITIONS: Rectal Cancer; Erectile Dysfunction
MeSH Terms: conditions — Rectal Neoplasms; Erectile Dysfunction | interventions — Laparoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Laparoscopic surgery (Sham Comparator): Patients receive no interventions after rectal cancer treatment.
  Interventions: Procedure: Laparoscopic surgery
- NeuroRegen scaffold transplantation (Experimental): Patients receive NeuroRegen scaffold transplantation after rectal cancer treatment.
  Interventions: Device: NeuroRegen scaffold transplantation
- NeuroRegen scaffold/BMMCs transplantation (Experimental): Patients receive autologous bone marrow mononuclear cells with NeuroRegen scaffold transplantation after rectal cancer treatment.
  Interventions: Biological: NeuroRegen scaffold/BMMCs transplantation
- NeuroRegen scaffold/HUC-MSCs transplantation (Experimental): Patients receive allogeneic human umbilical cord mesenchymal stem cells with NeuroRegen scaffold transplantation after rectal cancer treatment.
  Interventions: Biological: NeuroRegen scaffold/HUC-MSCs transplantation

INTERVENTIONS:
Procedure: Laparoscopic surgery — Completely resected rectal tumor.
  Arms: Laparoscopic surgery
Device: NeuroRegen scaffold transplantation — After completely resected rectal tumor, exposed pelvic autonomic nerves, and then transplanted NeuroRegen scaffold to the nerve.
  Arms: NeuroRegen scaffold transplantation
Biological: NeuroRegen scaffold/BMMCs transplantation — Completely resected rectal tumor, exposed pelvic autonomic nerves, and then transplanted NeuroRegen scaffold loaded with 5 million bone marrow mononuclear cells to the nerve.
  Arms: NeuroRegen scaffold/BMMCs transplantation
Biological: NeuroRegen scaffold/HUC-MSCs transplantation — Completely resected rectal tumor, exposed pelvic autonomic nerves, and then transplanted NeuroRegen scaffold loaded with 5 million human umbilical cord mesenchymal cells to the nerve.
  Arms: NeuroRegen scaffold/HUC-MSCs transplantation

SUMMARY:
Erectile dysfunction (ED) is one of the commonest complications in men after rectal cancer treatment. The purpose of this study is to assess the safety and efficacy of autologous bone marrow mononuclear cells (BMMCs) or allogeneic human umbilical cord-derived mesenchymal stem cells (HUC-MSCs) combined with NeuroRegen scaffold transplantation in men with erectile dysfunction after rectal cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with local rectal cancer, which is within 12cm from anus.
2. Male, 20-65 years old.
3. IIEF-5 score> 21.
4. No obvious abnormal in external genitalia, testis, epididymis and spermatic cord.
5. Have a consistent partner who is willing to engage in sexual activity more than twice per month during the study.
6. Signed informed consent.
7. Recently take no drugs affecting sexual function (such as androgen replacement drugs, PDE5i and Chinese patent medicine, etc.).

Exclusion Criteria:

1. Suffering hypertension or diabetes.
2. In the investigators judgment, with clinical significance of penis abnormalities, or has received penile prosthesis implantation surgery.
3. Patient's partner is trying to conceive during the trial period.
4. Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
5. Geographically inaccessible for follow-up visits required by protocol or want to other treatment.

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2016-01; Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Safety and Tolerability assessed by Adverse Events | Up to 6 months

SECONDARY OUTCOMES:
IIEF-5 (International Index of Erectile Function) | 1, 3, 6, 12 months
  Improvements in sexual function based on the (IIEF)-5 questionnaire
Mean scores of the Sexual Encounter Profile (SEP) Question 2, 3 | 1, 3, 6, 12 months
  Changes in mean scores of Sexual Encounter Profile (SEP) Question 2 and 3 will be evaluated and reported.
Penile cavernosal artery peak systolic velocity (PSV) | 1, 3, 6, 12 months
  Changes in penile cavernosal artery peak systolic velocity in [cm/s] as determined by Penile colour Doppler ultrasonography combined with prostaglandin-E1 injection.
Nocturnal penile tumescence (NPT) | 1, 3, 6, 12 months
  Monitor penis erection during sleep to assess erection function of the patients.
The change of results of Nerve electrophysiological examination | 1, 3, 6, 12 months
  To assess the penile sensory pathway abnormalities of the patients with or without premature ejaculation.
Maximum Flow Rate (Qmax) | 1, 3, 6, 12 months
  Change of the maximum flow rate (Qmax) to assess the bladder function.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D., Principal Investigator — Chinese Academy of Sciences
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China